CLINICAL TRIAL: NCT02839122
Title: A Study to Investigate the Pharmacokinetic Drug Interactions Between Dutasteride and Tadalafil in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuyu Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: YY_DUTA_2016
Record Dates: First submitted 2016-06-13; First posted 2016-07-20 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Benign Prostate Hyperplasia
Keywords: Dutasteride; Tadalafil
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil; Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dutasteride, Tadalafil (Experimental)
  Interventions: Drug: Tadalafil; Drug: Dutasteride
- Tadalafil, Dutasteride (Experimental)
  Interventions: Drug: Tadalafil; Drug: Dutasteride

INTERVENTIONS:
Drug: Tadalafil
Drug: Dutasteride

SUMMARY:
This is open-Label, A Randomized, Crossover study to evaluate the safety and pharmacokinetic interaction after oral concomitant administration of Dutasteride and Tadalafil in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 45 years
* BMI score 19 kg/m2 to 28 kg/m2
* SBP < 140 mmHg and ≤ 90 mmHg or DBP < 90 mmHg and ≥ 50 mmHg
* Eligible according to the laboratory results of hematology, blood chemistry and urinalysis
* Voluntarily signed the informed consent form

Exclusion Criteria:

* Gastrointestinal diseases or surgery which may affect absorption of the investigational products within 6 months
* History of hypersensitivity
* History of Cardiovascular disease
* History of degenerative Retina disease
* Lactose intolerance
* History of vision loss
* Clinically significant disorders of allergy, drug hypersensitivity reaction, hepatobiliary system, kidney, neurology, respiratory, hemato-oncology, endocrine, dermatology, urology, ophthalmology, psychiatry, musculo-skeletal system, immunology, otorhinolaryngology, and cardiovascular system
* Donated whole blood (transfusion, apheresis etc..) within 60 days
* Participated and administered the investigational products in other clinical trial within 90 days
* Taking drugs which may affect Clinical trial within 30 days
* Excessive alcohol consumption (> 3 units/week, 1 unit)
* Taking food which may affect Clinical trial within 7 days
* Positive result from Urinary test, Serum test
* Not eligible due to other reasons including laboratory results
* Clinically significant disorders result from Electrocardiography test
* Not eligible due to investigator's judgments

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve(AUC) of Dutasteride | 0,0.5,1,1.5,2,2.5,3,3.5,4,5,6,8,12,24,32,48,72,96,144,192,240 hours
Area Under the Curve(AUC) of Tadalafil, Dutasteride | 0,24,72,96,96.5,97,97.5,98,99,100,102,104,106,108,120,120.5,121,121.5,122,122.5,123,123.5,124,125,126,128,132,144,152,168,192,216,264,312,360 hours

CONTACTS AND LOCATIONS:
Overall Officials: hyeng-seok H Lim, ph.D, Principal Investigator — AIDS Malignancy Consortium

IPD SHARING:
Plan to Share IPD: Yes